CLINICAL TRIAL: NCT06849674
Title: Efficacy and Safety of Platelet-Rich Plasma as an Intraoperative Holding Solution in Hair Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, karem Taha ibrahim khalil, Assistant Professor of Dermatology,Venereology and Anddrology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP in hair transplantation
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hair Transplantation
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline group (Active Comparator): in this group, hair grafts will be stored in Normal saline 0.9% before transplantation.
  Interventions: Other: Saline
- Platelet-rich plasma group (Experimental): In this group, hair grafts will be stored in Platelet-rich plasma before transplantation.
  Interventions: Biological: Platelet rich plasma (PRP)

INTERVENTIONS:
Biological: Platelet rich plasma (PRP) — Hair grafts will be immersed in autologous Platelwt-richh plasma(PRP) before transplantation.
  Arms: Platelet-rich plasma group
Other: Saline — Hair grafts will be immersed in normal saline solution before transplantation.
  Arms: Saline group

SUMMARY:
The goal of this study is to determine the efficacy of using platelet-rich plasma (PRP) versus 0.9% normal saline as a storage solution during follicular unit extraction (FUE) hair transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male patients who have androgenetic alopecia
* Patients who are interested in having their hair transplanted

Exclusion Criteria:

* Individuals with comorbidities
* History of keloids or hypertrophic scarring
* Low donor area density
* Other causes of alopecia
* Scalp infections
* Patients with a bleeding tendency
* Patients on anticoagulant therapy
* Patients who are HIV-positive or Hepatitis B- or C-positive

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Change in Hair density | 12 weeks after hair transplantation
  Hair density (the number of hairs per square centimeter) will be measured using a trichoscope and digital photography in the recipient area.
Percentage of Hair Growth | 12 weeks after hair transplantation
  The percentage of graft survival will be assessed by comparing the number of transplanted hairs to the number of hairs that have grown in the recipient area using trichoscopic analysis and digital photography. The formula used will be: (number of grown hairs/number of transplanted hairs) x100%

SECONDARY OUTCOMES:
Patient satisfaction score | 12weeks after hair translantation
  Patient satisfaction will be assessed using Likert scale from 1 to 5 regarding aesthetic results, hair density, and natural appearance. Higher scores indicate greater satisfaction.
Incidence of Postoperative complications | within 1 month after hair transplantation
  The number and type of complications, including infection,graft necrosis, excessive shedding, and scalp irritation, will be documented. The severity of complications will be assessed using clinical examination and patient reports

CONTACTS AND LOCATIONS:
Overall Officials: Amany I Mustafa, MD, Study Director — Dermatology, Venereology and Andrology Faculty of Medicine- Benha University; Ahmed I Abdulkhaleq, MBBCh, Study Director — Dermatology, Venereology and Andrology Faculty of Medicine- Benha University
Locations (1):
- Dermatology, Venereology and Andrology Faculty of Medicine- Benha University, Banhā, Qalyubia Governorate, Egypt